CLINICAL TRIAL: NCT05163795
Title: Prediction of Fracture Nonunion Leading to Secondary Surgery in Patients With Distal Femur Fractures - Statistical Analysis Plan
Brief Title: Distal Femur Fracture Nonunion - Statistical Analysis Plan
Status: Completed | Type: Observational
Sponsor: Töölö Hospital (Other)
Responsible Party: Principal Investigator, Heini Sainio, Principal Investigator, Resident in Orthopedics and Traumatology, Töölö Hospital
Other Study IDs: Distal Femur Fractures - SAP
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Femur Distal Fracture; Nonunion of Fracture
Keywords: Prediction; Distal femur fracture; Nonunion; Statistical analysis plan
MeSH Terms: conditions — Femoral Fractures, Distal; Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lateral locking plate — Plating of the distal femur fracture with lateral locking plate.

SUMMARY:
Here the investigators describe the statistical analysis plan for the study assessing the prediction of fracture nonunion leading to secondary surgery in patients with distal femur fractures.

DETAILED DESCRIPTION:
See attached PDF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* AO/OTA type A or C distal femur fracture
* Fracture located on the metaphyseal area of the distal femur (square method)
* Operative treatment in the Helsinki University Hospital with a distal femur anatomic lateral locking plate
* Operative treatment within 1 month after trauma
* Operative treatment between years 2009 and 2018

Exclusion Criteria:

* Stress fracture
* Pathological fracture
* An epicondylar or subchondral fracture
* A ligament sprain in distal femur
* Treatment with a double-plating method or with both plate and nail
* Non-surgical treatment and patients who died before the treatment
* Treatment with an unconventional plate (other than distal femur plate)
* Patients whose follow-up criteria not fulfilled

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a retrospective cohort study conducted in level 1 trauma center at the Helsinki University Hospital with a catchment population of around one million for these fractures. All patients with a distal femur fracture treated at our institution between 2009 and 2018 were screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Reoperation | Within 36 months after the initial trauma
  Reoperation due to fracture nonunion

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lindahl, MD, PhD, Study Director — Department of Orthopaedics and Traumatology, University of Helsinki and Helsinki University Hospital, Helsinki, Finland
Locations (1):
- Department of Orthopaedics and Traumatology, University of Helsinki and Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication — https://boneandjoint.org.uk/Article/10.1302/2633-1462.48.BJO-2023-0077.R1

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT05163795/SAP_000.pdf